CLINICAL TRIAL: NCT02698436
Title: A Multi-Center, Evaluator Blinded, Randomized Clinical Study to Evaluate the Efficacy and Tolerance of Two Acne Treatments on Subjects With Mild to Moderate Acne Vulgaris
Brief Title: A Study to Evaluate the Effectiveness and Tolerance of Two Acne Treatments on Subjects With Mild to Moderate Acne.
Acronym: TIGER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CO-151211140520-SACT
Record Dates: First submitted 2016-02-26; First posted 2016-03-03 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Acne Vulgaris
Keywords: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Acne Mask (Experimental): The light therapy acne device is applied to the face once in the evening for a duration of 10 minutes. The cleanser is used twice daily, once in the morning and once in the evening.
  Other Names: Cleanser is marketed while the device is not marketed
  Interventions: Device: Acne Mask
- 2.5% Benzoyl Peroxide Treatment (Active Comparator): Cleanser and 2.5% Benzoyl Peroxide Treatment Both the cleanser and the 2.5% Benzoyl Peroxide Treatment are applied twice daily, once in the morning and once in the evening.
  Other names: Both products are marketed
  Interventions: Drug: 2.5% Benzoyl Peroxide Treatment

INTERVENTIONS:
Device: Acne Mask — The light therapy device contains a combination of red and blue light-emitting diodes. The device is applied once daily, in the evening for a duration of 10 minutes
  Other Names: Light-Therapy Acne Device
  Arms: Acne Mask
Drug: 2.5% Benzoyl Peroxide Treatment — The BPO treatment is applied twice daily, once in the morning and once in the evening
  Other Names: BPO
  Arms: 2.5% Benzoyl Peroxide Treatment

SUMMARY:
This study will compare two different acne treatments for the treatment of acne. Half of the participants will receive two marketed acne products (cleanser and leave-on topical treatment), while the other half of the participants will receive a marketed cleanser and a light-therapy device.

DETAILED DESCRIPTION:
Acne is a common chronic skin disease involving blockage and/or inflammation of the hair follicles and their accompanying sebaceous gland.

Benzoyl peroxide (BPO) is one of the most effective and well-studied over-the-counter (OTC) acne therapies, is generally regarded as safe and effective and is considered as a first-line treatment for acne. Topical BPO monotherapy products for at-home acne treatment have been available for OTC use for more than 30 years and studies have indicated that a low dose of BPO may be an effective approach for treating acne using an OTC product when applied consistently to larger areas of the face due primarily to its effects against acne-causing bacteria.

BPO has anti-inflammatory and keratolytic properties, but is thought to act primarily to control P. acnes by releasing reactive oxygen species that are toxic to the bacteria. The most common side effect of topical BPO treatment is skin irritation, which can include erythema, burning, and peeling.

As an alternative to topical OTC standard of care therapies, research has also shown the benefits of red and blue light therapy in the treatment of mild to moderate acne, with red and blue light shown to target the acne-causing bacteria and have an effect on inflammation reduction.

Light-based therapies have been successfully used to treat dermatological conditions since the early 1900's, with various parts of the electromagnetic spectrum (i.e. UV, visible, near-Infrared, etc.) demonstrating different benefits. Light-emitting diodes (LEDs) offer delivery of light to the skin in a gentler manner as compared to light delivered by lasers primarily due to the lower energy output. It has been reported that LEDs do not deliver enough power to damage tissues and do not have the same risk of accidental eye damage that lasers do. Visible-LED light therapy has been deemed a non-significant risk by the Food and Drug Administration and has been approved for use in humans.

This study will look to compare the acne clearing efficacy and tolerance of two different acne treatments: a currently marketed 2.5% BPO full-face topical OTC treatment, and an Investigational red and blue light acne light therapy mask, to determine if the acne resolution efficacy of the Investigational mask is as effective as a current OTC standard of care for at-home treatment of mild to moderate acne.

ELIGIBILITY:
Inclusion Criteria:

* Has mild to moderate acne
* Has 10 - 100 pimples, 10 - 50 inflamed red pimples, up to 2 raised bumps and no cysts
* In general good health
* Must avoid excessive sun exposure and any light treatments or any professional or aesthetic spa-like procedures
* Must not be pregnant, nursing or intend to become pregnant during the study
* Must agree to practice a medically acceptable form of birth control.
* Must be able to read, speak, write and understand English

Exclusion Criteria:

* Allergies or sensitivities to product ingredients or to light
* Has severe acne or pre-existing dermatological facial condition
* Has an uncontrolled disease or immune deficient disorder
* Is pregnant, breast-feeding or intending to become pregnant
* Has been taking prescription drug medication for acne or antibiotics for the past 6 months

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 103 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alicia D Bucko, D.O., Principal Investigator — Academic Dermatology Associates; Lily Jiang, Ph.D., Principal Investigator — Thomas J. Stephens and Associates, Inc.
Locations (2):
- United States (2):
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Thomas J. Stephens and Associates, Inc., Richardson, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ashkenazi H, Malik Z, Harth Y, Nitzan Y. Eradication of Propionibacterium acnes by its endogenic porphyrins after illumination with high intensity blue light. FEMS Immunol Med Microbiol. 2003 Jan 21;35(1):17-24. doi: 10.1111/j.1574-695X.2003.tb00644.x. PMID 12589953
- [Background] Kjeldstad B. Photoinactivation of Propionibacterium acnes by near-ultraviolet light. Z Naturforsch C Biosci. 1984 Mar-Apr;39(3-4):300-2. doi: 10.1515/znc-1984-3-417. PMID 6730638
- [Background] Barolet D. Light-emitting diodes (LEDs) in dermatology. Semin Cutan Med Surg. 2008 Dec;27(4):227-38. doi: 10.1016/j.sder.2008.08.003. PMID 19150294

RESULTS

PARTICIPANT FLOW:
Groups:
- Acne Mask: Light therapy mask applied to the face once in the evening for a duration of 10 minutes
- Benzoyl Peroxide 2.5%: Apply test product to face once in the morning and once at night.
Period: Overall Study
Arm/Group | Acne Mask | Benzoyl Peroxide 2.5%
Started | 59 | 58
Completed | 52 | 51
Not Completed | 7 | 7
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Lost to Follow-up | 2 | 4
Not completed — Non-compliance with study regimen | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- 2.5% Benzoyl Peroxide Treatment: Applied BPO treatment once daily
- Total: Total of all reporting groups
Arm/Group | Acne Mask | 2.5% Benzoyl Peroxide Treatment | Total
Number analyzed (Participants) | 59 | 58 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.8 (5.79) | 18.7 (5.97) | 18.2 (5.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 | 62
  Male | 28 | 27 | 55
Region of Enrollment [Number; unit: participants]
  USA | 59 | 58 | 117

OUTCOME MEASURES:

1. Primary Outcome: Percent Change of Global Face Total Acne Lesion Count From Baseline
Time Frame: Baseline to 12 Weeks
Population: Includes all subjects who had measurements taken at this time point. Some subjects may have missed the visit, or had a protocol deviation that would exclude their data.
Measure: Mean (95% Confidence Interval); unit: Percent change of acne lesion count
Groups:
- 2.5% Benzoyl Peroxide: Both 2.5% BPO cleanser and treatment are applied twice daily, once in the moring and once in the evening
Arm/Group | Acne Mask | 2.5% Benzoyl Peroxide
Number analyzed (Participants) | 55 | 54
Percent change of acne lesion count | -44 [-51 to -37] | -54 [-61 to -45]

2. Secondary Outcome: Percent Change of Global Face Total Acne Lesion Count From Baseline to Week 1
Time Frame: Baseline to 1 Week
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percent change of acne lesion count
Arm/Group | Acne Mask | 2.5% Benzoyl Peroxide
Number analyzed (Participants) | 54 | 54
Percent change of acne lesion count | -19 [-25 to -13] | -26 [-33 to -19]

3. Secondary Outcome: Percent Change of Global Face Total Acne Lesion Count From Baseline to Week 2
Time Frame: Baseline to 2 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percent change of acne lesion count
Arm/Group | Acne Mask | 2.5% Benzoyl Peroxide
Number analyzed (Participants) | 52 | 52
Percent change of acne lesion count | -28 [-35 to -21] | -42 [-48 to -35]

4. Secondary Outcome: Percent Change of Global Face Total Acne Lesion Count From Baseline to Week 4
Time Frame: Baseline to 4 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percent change of acne lesion count
Arm/Group | Acne Mask | 2.5% Benzoyl Peroxide
Number analyzed (Participants) | 54 | 52
Percent change of acne lesion count | -35 [-42 to -27] | -46 [-53 to -39]

5. Secondary Outcome: Percent Change of Global Face Total Acne Lesion Count From Baseline to Week 8
Time Frame: Baseline to 8 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percent change of acne lesion count
Arm/Group | Acne Mask | 2.5% Benzoyl Peroxide
Number analyzed (Participants) | 52 | 51
Percent change of acne lesion count | -40 [-46 to -33] | -50 [-62 to -38]

6. Secondary Outcome: Acne Lesion Counts Total Global Face - Baseline
Description: Acne Lesion Count Total Global Face at Baseline
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Lesion Count
Arm/Group | Acne Mask | 2.5% Benzoyl Peroxide
Number analyzed (Participants) | 55 | 54
Lesion Count | 47.2 (22.56) | 47.6 (23.22)

7. Secondary Outcome: Acne Lesion Counts Total Global Face - Week 1
Description: Acne Lesion Count Total Global Face Week 1
Time Frame: 1 Week
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Lesion Count
Arm/Group | Acne Mask | 2.5% Benzoyl Peroxide
Number analyzed (Participants) | 54 | 54
Lesion Count | 39.2 (22.5) | 36.8 (24.00)

8. Secondary Outcome: Acne Lesion Counts Total Global Face - Week 2
Description: Acne Lesion Count Total Global Face Week 2
Time Frame: 2 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Lesion Count
Arm/Group | Acne Mask | 2.5% Benzoyl Peroxide
Number analyzed (Participants) | 52 | 52
Lesion Count | 35.3 (20.13) | 30.5 (22.88)

9. Secondary Outcome: Acne Lesion Counts Total Global Face - Week 4
Description: Acne Lesion Count Total Global Face Week 4
Time Frame: 4 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Lesion Count
Arm/Group | Acne Mask | 2.5% Benzoyl Peroxide
Number analyzed (Participants) | 54 | 52
Lesion Count | 30.5 (17.51) | 27.0 (19.76)

10. Secondary Outcome: Acne Lesion Counts Total Global Face - Week 8
Description: Acne Lesion Count Total Global Face Week 8
Time Frame: 8 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Lesion Count
Arm/Group | Acne Mask | 2.5% Benzoyl Peroxide
Number analyzed (Participants) | 52 | 51
Lesion Count | 27.8 (16.06) | 26.4 (28.40)

11. Secondary Outcome: Acne Lesion Counts Total Global Face - Week 12
Description: Acne Lesion Count Total Global Face Week 12
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Lesion Count
Arm/Group | Acne Mask | 2.5% Benzoyl Peroxide
Number analyzed (Participants) | 52 | 51
Lesion Count | 24.8 (15.76) | 23.3 (20.91)

12. Secondary Outcome: Investigator Global Acne Assessment - Baseline
Description: Investigator's assessment of subject's acne condition using a score of 0 (best) and 5 (worst) on the Modified Cook's scale.
  0 Clear Residual hyperpigmentation and erythema may be present.
  1. Almost Clear. A few scattered comedones and a few (less than five) small papules.
  2. Mild.Easily recognizable; less than half the face is involved. Many comedones and many papules and pustules.
  3. Moderate More than half of the face is involved. Numerous comedones, papules and pustules.
  4. Severe. Entire face is involved. Covered with comedones, numerous papules and pustules and few nodules and cysts.
  5. Very Severe.Highly inflammatory acne covering the face; with nodules and cysts present.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Acne Mask | 2.5% Benzoyl Peroxide
Number analyzed (Participants) | 55 | 54
Score on a scale | 2.55 (0.529) | 2.51 (0.471)

13. Secondary Outcome: Investigator Global Acne Assessment - Week 1
Description: as for outcome 12
Time Frame: 1 Week
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Acne Mask | 2.5% Benzoyl Peroxide
Number analyzed (Participants) | 54 | 54
Score on a scale | 2.35 (0.538) | 2.34 (0.548)

14. Secondary Outcome: Investigator Global Acne Assessment - Week 2
Description: as for outcome 12
Time Frame: 2 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Acne Mask | 2.5% Benzoyl Peroxide
Number analyzed (Participants) | 52 | 52
Score on a scale | 2.23 (0.598) | 2.11 (0.605)

15. Secondary Outcome: Investigator Global Acne Assessment - Week 4
Description: as for outcome 12
Time Frame: 4 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Acne Mask | 2.5% Benzoyl Peroxide
Number analyzed (Participants) | 54 | 52
Score on a scale | 2.08 (0.612) | 1.87 (0.650)

16. Secondary Outcome: Investigator Global Acne Assessment - Week 8
Description: as for outcome 12
Time Frame: 8 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Acne Mask | 2.5% Benzoyl Peroxide
Number analyzed (Participants) | 52 | 51
Score on a scale | 1.88 (0.583) | 1.70 (0.775)

17. Secondary Outcome: Investigator Global Acne Assessment - Week 12
Description: as for outcome 12
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Acne Mask | 2.5% Benzoyl Peroxide
Number analyzed (Participants) | 52 | 51
Score on a scale | 1.77 (0.660) | 1.59 (0.726)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the informed consent/assent was obtained through the subject's last study procedure/visit. Serious adverse events were also collected 30 calendar days beyond the subject's last procedure/visit and longer if study-related.
Arm/Group | Acne Mask | 2.5% Benzoyl Peroxide Treatment
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/58
Other Adverse Events (participants affected / at risk) | 0/59 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No